CLINICAL TRIAL: NCT01753882
Title: Monoaminergic Modulation of Motor Function in Subacute Incomplete Spinal Cord Injury
Brief Title: Monoaminergic Modulation of Motor Function in Subacute Incomplete Spinal Cord Injury (SCI)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Thomas G Hornby, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00056589
Record Dates: First submitted 2012-12-06; First posted 2012-12-20 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Spinal Cord Injury
Keywords: Gait training; Lexapro; Tizanidine
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gait Training with Lexapro (Experimental): Gait training 2 weeks, gait training for 4 weeks (3X week) with Lexapro (10 mg SSRI), wash out period of 1 week, gait training for 4 weeks with placebo (10 mg). Patients will also be provided prescribed TIZ by their physician to help control of spastic motor behaviors.
  Interventions: Drug: Lexapro
- Gait Training with Placebo (Active Comparator): Gait training 2 weeks, gait training for 4 weeks (3X week) with Placebo (10 mg), wash out period of 1 week, gait training for 4 weeks with Lexapro(10 mg). Patients will also be provided prescribed TIZ by their physician to help control of spastic motor behaviors.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lexapro — Agent + training vs Placebo + training
  Other Names: escitalopram
  Arms: Gait Training with Lexapro
Drug: Placebo — Agent + training vs Placebo + training
  Other Names: microcrystalline dextrose
  Arms: Gait Training with Placebo

SUMMARY:
The primary goal of the proposed clinical trial is to investigate the combined effects of walking training and monoaminergic agents (SSRIs and TIZ) on motor function of individuals in sub-acute (2-7 mo) human motor incomplete Spinal Cord Injury (SCI), with a primary emphasis on improvement in locomotor capability. We hypothesize that the use of these drugs applied early following SCI may facilitate independent stepping ability, and its combination with intensive stepping training will result in improved locomotor recovery following incomplete SCI. Loss of descending control via norepinephrine inputs following spinal cord injury can impair normal sensorimotor function through depressing motor excitability and impairing walking capacity. Replacing these inputs with drugs can alter the excitability and assist with reorganization of locomotor circuits. Assessment of single-dose administration of these agents has been tested in patients with motor incomplete spinal cord injury; only limited changes in walking performance have been noted. The resultant onset of weakness and increase in involuntary reflexes following motor incomplete SCI may partly be a result of damage to descending pathways to the spinal cord that control the release of serotonin. In models of SCI, for example, application of agents that simulate serotonin has been shown to change voluntary motor behaviors, including improvement of walking recovery. In humans following neurological injury, the effects of 5HT agents are unclear. Few previous reports indicate improved motor function following administration of agents which enhance the available serotonin in the brain, although some data suggests that increased serotonin may be beneficial. In this application, we propose to study the effects of clinically used agents that increase or decrease intrinsic serotonin activity in the brain on strength and walking ability following human motor incomplete SCI. Using detailed electrophysiological recordings, and biomechanical and behavioral measures, we will determine the effects of single or chronic doses of these drugs on voluntary and involuntary motor behaviors during clinical measures and walking measures. The novelty of this proposed research is the expectation that agents that increase serotonin activity may increase abnormal reflexes in SCI, but simultaneously help to facilitate motor and walking recovery. Despite potential improvements in voluntary function, the use of pharmacological agents that may enhance spastic motor behaviors following SCI is in marked contrast to the way in which drugs are typically used in the clinical setting.

DETAILED DESCRIPTION:
This is a phase I double blinded randomized control clinical trial. The procedures for participation in both Aims of the study are described below in chronological order.

Aim 1 and 2: Explanation of the consent form and study procedures/protocol will be performed in the Neurolocomotion laboratory (room 1382), with subjects and their families provided ample time for questions. Subjects are provided substantial time to choose to participate, and are provided the laboratory phone numbers/emails to contact the PI and research personnel with any potential questions. In situations where the subject is unable to be transported to the laboratory, the PI will explain the consent form at a time and location convenient for the subject and/or their family. Subjects will then undergo a screening procedure to determine if they are eligible to participate in the study based on inclusion/exclusion criteria.

Aim 1:

Modified Ashworth scale (mod Ash, no units) will be used to detect velocity-dependent resistance to passive muscle stretch/joint rotation. The modAsh will grossly assess spasticity at bilateral knee extensors and knee flexors, with scores from 0-5 (1+ scores will be converted to 2 and higher scores increased accordingly).

Spinal Cord Assessment Tools for Spasticity (SCATS, no units) will be employed to assess flexor and extensor spasms and clonic activity of the plantarflexors (Benz et al. , 2005).

Independence in walking ability will be assessed at each assessment period using the Walking Index for SCI II (WISCI II, which is a 21 point (0-20) ordinal scale which assigns a score based on amount of physical assistance, bracing, and assistive device used to ambulate. Notably, subjects will not be allowed to ambulate with braces extending above the knee. Six minute walk test (m) will be assess walking around a continuous hall-way at subjects' self-selected velocity, with distance determined each minute and summed over the entire six minute duration (van Hedel et al. , 2005). Subjects will be asked to "walk at your (their) normal, comfortable pace" with minimal physical assistance and bracing/devices as needed This measure is significantly association with measures of community walking in subjects with incomplete SCI (Saraf et al. , 2009).

BERG balance test will be administered. Gait Mat testing will be performed to guage spatiotemporal aspects of walking. 6 minute walk test will be performed. Lower Extremity Motor Score, Peak treadmill speed (m/s)

Aim 2:

Same as above including strength evaluations : Ankle, knee, hip flexors/extensors tested bilaterally (Biodex®).

Subjects in Aim 2 will be tested at initial evaluation, after four weeks of initial training, and will be repeated after each four weeks of training on either the placebo or study medication.

Subjects in Aim 2 will additionally be requested to return for follow up testing after one year.

Subjects will be offered to participate in audio, videotaping and/or photography.

Women who are of childbearing age and are contemplating becoming pregnant will be required to submit a pregnancy test and must notify the principal investigator immediately.

ELIGIBILITY:
Inclusion Criteria:

A) Subjects with motor incomplete SCI (AIS C or D) of 1-9 mo. duration will be selected, with anatomical lesions between C1-T10.

B) Subjects will be between 18 and 75 years of age . Note: grant application states 16-75, however, we will be only including subjects 18-75.

C) All subjects must be previously ambulatory with passive range of motion consistent with normal walking, and must include: ankle dorsiflexion ankle to 10° and plantarflexion to 30°, knee flexion from 0 to 90°, hip flexion/extension to 90° - -10°.

D) Subjects will be medically stable with medical clearance to participate, with absence of concurrent severe medical illness, including unhealed decubiti, existing infection, significant cardiovascular or metabolic disease which limits exercise participation, significant osteoporosis (as indicated by history of fractures following injury), active heterotrophic ossification in the lower extremities, known history of peripheral nerve injury in lower legs, history of known traumatic head injury, and history of pulmonary complications, including significant obstructive and/or restrictive lung diseases.

E) Individuals who are undergoing concurrent physical therapy will not be excluded from the study population, secondary to the use of the cross-over design. Physical therapy records will be obtained to ascertain the amount and types of physical therapy services being provided.

F) Women of childbearing potential will not be excluded, although women who are pregnant or who are considering becoming pregnant will be excluded due to the trunk and pelvis restraints required for use during locomotion, and secondary to the unknown effects of the pharmacological agents on the developing fetus.

G) Patients with known liver, renal, or other metabolic disease that may interfere with drug action and/or clearance will be excluded from the proposed study. These complications will be partially obviated by requiring all patients to undergo specific medical procedures (liver function tests, urinalysis) prior to admission.

H)Men and women will be recruited for participation in the proposed clinical trial at rates consistent with national and local average of gender disparities of SCI (80% male, 20% women). Women of childbearing potential will not be excluded, although women who are pregnant or who are considering becoming pregnant will be excluded due to the trunk and pelvis restraints required for use during locomotion, and secondary to the unknown effects of the test agent (SSRIs) on the developing fetus. Women who use oral contraceptives will not be assessed for TIZ experiments and will be excluded from Aim 1.

I) Individuals of different ethnicities will be recruited at rates similar to the national and local ethnicity rates. Current data since 2005 indicate that of the entire population of SCI, 66.1% are Caucasian, 27.1% are African American, 6.6% are of Hispanic origin, and 2.0% are Asian. These populations closely resemble those at RIC and in our previous studies in human SCI.

Exclusion Criteria:

A) Subjects who are ventilator-dependent will be excluded secondary to severely impaired respiratory capacity.

B) Subjects with substantial orthopedic bracing to stabilize the cervical or thoracic vertebral column and are unable to fit in the safety harness without increased risk of injury are not eligible.

C) Patients will also be excluded if they are unable to tolerate 10 minutes of standing without orthostasis (decrease in blood pressure by 20 mmHg systolic and 10 mmHg diastolic); previous experience in the sub-acute population suggests that 10 minutes of standing is more than sufficient for tolerating 45 minutes of walking secondary to increased activity/muscle pump minimizing risk for orthostasis.

D) Women who are pregnant or who are considering becoming pregnant will be excluded due to the trunk and pelvis restraints required for use during locomotion, and secondary to the unknown effects of the pharmacological agents on the developing fetus.

E) Subjects with height and weight limitations which restrict participation in Lokomat Training(LT) will be excluded. For height, subjects who are > 78 inches or < 60 inches tall may present with thigh/shank lengths that may limit use of the Lokomat. If subjects are not able to step independently on the treadmill and require use of robotic-assistance during treadmill stepping, attempts to fit all subjects in the robotic orthosis prior to enrollment and randomization. For weight, the maximum weight limit for use of the safety harness/counterweight system is 300 lbs.

F) Individuals with concurrent severe medical illness, including unhealed decubiti, existing infection, significant cardiovascular or metabolic disease which limits exercise participation, significant osteoporosis (as indicated by history of fractures following injury), active heterotrophic ossification in the lower extremities, known history of peripheral nerve injury in lower legs, history of known traumatic head injury, and history of pulmonary complications, including significant obstructive and/or restrictive lung diseases will be excluded.

G) Patients prescribed other anti-depressant medications, including specific monoaminergic agents, their precursors or their agonists, or other medications with known interactions to the SSRIs or TIZ will be excluded. With consultation and supervision of the patients' physician and the attending physicians for each individual patient, subjects will be required to wean of their medications on an appropriate and safe dosing schedule to minimize side effects of drug cessation or withdrawal. All subjects will be excluded from participation unless both attending physician and patient agree to cease all such medications during the evaluation and training period. A 14-day washout period for SSRIs and a 72 hour washout for TIZ will be utilized.

H) All subjects prescribed anti-spastic medications will be excluded. Specific agents to be excluded include baclofen (Lioresal®) and benzodiazepines (Diazepam®). Selected agents used for pain modulation will be evaluated per subject to ascertain potential interactions with test agent. With consultation and supervision of the patients' physician and the attending physicians for each individual patient, subjects will be required to wean of their medications on an appropriate and safe dosing schedule to minimize side effects of drug cessation or withdrawal. All subjects will be excluded from participation unless both attending physician and patient agree to cease all such medications during the evaluation and training period. A 72-hour minimum washout period for all such medications will be utilized. (Note: exception to use of TIZ during training - see above).

I) Women of childbearing potential will not be excluded, although women who are pregnant or who are considering becoming pregnant will be excluded due to the trunk and pelvis restraints required for use during locomotion, and secondary to the unknown effects of the test agent (SSRIs) on the developing fetus. Women who use oral contraceptives will not be assessed for TIZ experiments and will be excluded from Aim 1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2012-02; Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Walking Index for Spinal Cord Injury (WISCI II) | Compare changes in WISCI II pre to post training with placebo to pre to post training with Lexapro during a 10-12 week time period.
  Evaluation of bracing, assistive device, and assistance required for ambulation
Peak treadmill velocity | Compare changes in peak treadmill velocity pre to post training with placebo to pre to post training with Lexapro during a 10-12 week time period.
  During graded treadmill test

SECONDARY OUTCOMES:
Volitional Strength | Pre Training (Day 1), Pre Drug B (approx end of week 5), Post-Final (approx end of week 10)
  Ankle, knee, hip flexors/extensors strength (Nm) tested bilaterally (Biodex®)
Gait kinematics | Pre Training (Day 1), Pre Drug A (approx end of week 2), Post Drug A (approx end of week 4), Pre Drug B (approx end of week 5), Post Drug B (approx end of week 9), Post-Final (approx end of week 10)
  Kinematic excursions of hip/knee/ankle (Motion Analysis®)
Fastest possible walking velocity over ground (FV; m/s) | Pre Training (Day 1), Pre Drug A (approx end of week 2), Post Drug A (approx end of week 4), Pre Drug B (approx end of week 5), Post Drug B (approx end of week 9), Post-Final (approx end of week 10)
  Subject walks a distance of 10m with the middle 6m being timed. Instructions to walk normal comfortable pace.
Six minute walking distance (m) | Pre Training (Day 1), Pre Drug A (approx end of week 2), Post Drug A (approx end of week 4), Pre Drug B (approx end of week 5), Post Drug B (approx end of week 9), Post-Final (approx end of week 10)
  Subject asked to walk normal comfortable pace for 6 minutes. Total distance is recorded. Subject can take rest breaks as needed but are encouraged to continue walking throughout the 6 minutes.
Lower Extremity Motor Scores (LEMS) | Pre Training (Day 1), Pre Drug A (approx end of week 2), Post Drug A (approx end of week 4), Pre Drug B (approx end of week 5), Post Drug B (approx end of week 9), Post-Final (approx end of week 10)
  Measure of lower extremity muscle strength on 0-5 point scale.
Modified Ashworth of knee extensors/flexors (modAsh) | Pre Training (Day 1), Pre Drug A (approx end of week 2), Post Drug A (approx end of week 4), Pre Drug B (approx end of week 5), Post Drug B (approx end of week 9), Post-Final (approx end of week 10)
  Measure of spasticity of knee flexors and extensors during passive range of motion
Spinal Cord Assessment Tool for Spasticity (SCATS) | Pre Training (Day 1), Pre Drug A (approx end of week 2), Post Drug A (approx end of week 4), Pre Drug B (approx end of week 5), Post Drug B (approx end of week 9), Post-Final (approx end of week 10)
  Measure of spasticity tested in supine

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States